CLINICAL TRIAL: NCT06034691
Title: Exploratory Research of PCSK9 Inhibitor on Patency of Autogenous Arteriovenous Fistula After Percutaneous Transluminal Angioplasty With Paclitaxel Releasing Balloon
Brief Title: Exploratory Research of PCSK9 Inhibitor on Patency of aAVF After PTA With PCB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LY2023-113-A
Record Dates: First submitted 2023-08-14; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Hemodialysis Access Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCSK9i group (Experimental): treatment group
  Interventions: Biological: pcsk9 inhibitor
- control group (No Intervention): control group

INTERVENTIONS:
Biological: pcsk9 inhibitor — The treatment group received postoperative use of 140 mg of Ribavirin, administered every two weeks, with 140 mg administered subcutaneously for a total of 48 weeks. There was no additional intervention with lipid-lowering drugs in the control group.
  Arms: PCSK9i group

SUMMARY:
Autologous arteriovenous fistula (AVF) is the preferred vascular pathway type for maintenance hemodialysis (MHD) patients. The K/DOQI guidelines suggest that the use of percutaneous transluminal angioplasty (PTA) as the primary treatment for AVF stenosis is reasonable. However, the durability of PTA is limited. In order to reduce the risk of dysfunction recurrence after the intervention, there have been reports in recent years that drug-coated balloons (DCB) are used in the treatment of vascular stenosis in hemodialysis. Multiple factors have limited the efficacy of DCB. Previous studies on the related factors of hemodialysis access stenosis showed that Dyslipidemia was significantly related to the short initial patency rate, and Dyslipidemia was an important predictor of secondary patency loss. Proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors are a new type of lipid-lowering drug that can prevent vascular calcification. Previous studies have shown that PCSK9 inhibitors have good lipid-lowering effects in both MHD patients and nondialysis patients, and the use of PSK9 inhibitors at the same dose as nondialysis patients is safe in MHD patients. There are currently few studies on the use of paclitaxel-releasing balloon dilation combined with PCSK9 inhibitors to improve autologous internal fistula. Therefore, the investigators applied a prospective, randomized, and controlled study method to preliminarily explore the effect of paclitaxel releasing balloon combined with PCSK9 inhibitor on improving the postoperative patency rate of AVF and the safety of the combined application.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to join this study and sign an informed consent form
2. Age ≥ 18 years old and ≤ 75 years old, regardless of gender
3. Maintenance hemodialysis patients using autologous arteriovenous fistula (AVF), with a dialysis frequency of three times a week
4. AVF venous stenosis: The local stenosis rate exceeds 50% of the normal diameter of nearby blood vessels and is accompanied by at least one of the following conditions:

   1. The natural blood flow of the internal fistula is less than 500ml/min or has decreased by more than 25% compared to the previous examination result
   2. Unable to meet the required blood flow for dialysis prescription (blood flow<200ml/min, and cannot be corrected after adjusting the puncture needle position)
   3. Decreased arterial pressure or increased venous pressure during dialysis (monitoring arterial pressure<-120mmHg for more than 2 consecutive times or monitoring venous pressure>120mmHg while maintaining 200ml/min blood flow)
   4. Difficulty in puncture: A qualified nurse who has difficulty puncturing for 3 consecutive days of hemodialysis (blood can only be drawn out after more than two punctures)
   5. Decreased dialysis adequacy [arteriovenous fistula recirculation rate (RA)>10%, or an increase of more than 25% compared to the previous examination result] [RA=(SA-A)/(SA-V) * 100, dialysis to 1 hour: SA=blood flow adjusted to 20ml/min, ultrafiltration and dialysate flow stopped, after 2 minutes, artery Blood urea nitrogen concentration A=artery Blood urea nitrogen concentration V=vein Blood urea nitrogen concentration]
   6. Abnormal signs of fistula.
5. Patients with primary Hypercholesterolemia [LDL-C ≥ 130 mg/dl (≥ 3.4 mmol/L), and/or non-HDL-C≥ 160 mg/dl (≥ 4.1 mmol/L)] or combine cardiovascular disease or assess patients with a high risk of cardiovascular disease

Exclusion Criteria:

1. MHD with AVG
2. Breastfeeding or Pregnant Women
3. Patients with central venous reflux obstruction
4. Patients with AVF feeding artery disease
5. Patients with severe Hypotension (systolic blood pressure<90mmHg or diastolic blood pressure<60mmHg, at least three times within one month before signing the informed consent)
6. Left ventricular Ejection fraction less than 30% or hemodynamic instability
7. Patients receiving immunotherapy or suspected/confirmed Vasculitis
8. Patients with coagulation dysfunction or a history of Thrombocytopenic purpura
9. Patients with vascular access infections or systemic active infections
10. Patients who are known to be allergic to PCSK9 inhibitors or paclitaxel
11. Patient's life expectancy is less than 12 months
12. Patients who are planning kidney transplantation or switching to Peritoneal dialysis
13. Patients participating in other intervention studies
14. The researcher judged that the subject's condition was not suitable for participation in this study

Ages: 17 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2024-09-06 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Value of vessel diameter | 24 week, 48 week
  ultrasonic measurement
Value of volume of blood flow | 24 week, 48 week
  ultrasonic measurement
Value of peak systolic velocity ratio（PSVR） | 24 week, 48 week
  ultrasonic measurement
Incidence of Re intervention of fistula | 48 week
  Event recording

SECONDARY OUTCOMES:
Endometrium | 24 week, 48 week
  Ultrasonic measurement of changes in thickness of vascular intima , expressed in millimeters
RA | 24 week, 48 week
  Arteriovenous fistula recirculation rate
BTM | 24 week, 48 week
  Blood temperature monitoring, testing of specific modules of the hemodialysis machine. Expressed as a percentage.
Adequacy of dialysis | 24 week, 48 week
  spKT/V
Blood routine | 12 week, 24 week, 48 week
  Concentration of hemoglobin, white blood cell count, platelet
liver function | 12 week, 24 week, 48 week
  Concentration of GPT, GOT
Concentration of blood sugar | 12 week, 24 week, 48 week
Concentration of CRP | 12 week, 24 week, 48 week
blood lipids | 12 week, 24 week, 48 week
  Concentration of cholesterol, triglyceride, LDL-c, HDL

CONTACTS AND LOCATIONS:
Locations (1):
- Yuanyuan Xie, Shanghai, Pudong, China